CLINICAL TRIAL: NCT04777422
Title: A Pilot Study to Determine the Safety of Defibrotide in Children With High Risk Kawasaki Disease
Brief Title: Defibrotide in Children With High Risk Kawasaki Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Medical College (Other)
Collaborators: Johns Hopkins University (Other); Columbia University (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-204
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki; Children; Defibrotide
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Defibrotide 6.25 mg/kg IV q6h
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide 6.25 mg/kg IV q6h up to 7 days
  Other Names: Defitelio®

SUMMARY:
This study evaluates the safety of defibrotide with IVIG in children with high risk Kawasaki disease.

ELIGIBILITY:
Inclusion Criteria:

* Kawasaki disease presumptive diagnosis defined according AHA criteria;
* Signed informed consent and patient assent (if applicable)
* Diagnosis of KD and initiation of defibrotide within 96 hours from the conclusion of IVIG treatment
* Age: 0 - 11 years old
* High risk category defined as patient meeting ≥2 of the following criteria: male, age <6 months or >8yrs, IVIG-resistance, Fever lasting greater than 10 days, prior to diagnosis, Coronary artery aneurysms, and/or Laboratory tests indicating worse systemic inflammation
* PT and PTT within institutional normal limits
* Platelet count ≥100,000/mm3

Exclusion Criteria:

* History of Grade III or IV hemorrhage or active bleeding;
* Previous Grade II-IV hypersensitivity to defibrotide
* Current systemic anti-coagulant therapy and/or fibrinolytic therapy, excluding aspirin (5 mg/kg/dose maximum).
* Patients on an active experimental trial for Kawasaki disease

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with grade III/IV allergic reaction to defibrotide | 30 days
  All patients will be monitored for allergic reaction probably or definitely related to defibrotide administration.
Number of patients with grade III/IV hemorrhage attributable to defibrotide | 42 days
  All patients will be monitored for hemorrhage probably or definitely related to defibrotide.

SECONDARY OUTCOMES:
Number of patients with improvement in clinical progression/signs of Kawasaki disease | 42 days
  Patients will have pre and post treatment assessments with imaging and blood tests to monitor clinical signs of Kawasaki disease

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Cairo, MD, Principal Investigator — New York Medical College
Locations (3):
- United States (3):
  - Columbia University, New York, New York
  - New York University, New York, New York
  - Mitchell Cairo, Valhalla, New York